CLINICAL TRIAL: NCT06702384
Title: A Prospective Translational Tissue Collection Study in Early and Advanced Gastric and Oesophageal Cancers to Enable Further Disease Characterisation and the Development of Potential Predictive and Prognostic Biomarkers
Brief Title: Molecular Analysis of Gastric and OEsophageal Cancers STudy
Acronym: MAGnET
Status: Withdrawn | Type: Observational
Why Stopped: Never opened to recruitment due to lack of funding
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 5139; 20/LO/0506 (Other: REC reference); 264017 (Other: IRAS project ID)
Record Dates: First submitted 2022-02-24; First posted 2024-11-25 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-09

CONDITIONS: Adenocarcinoma Esophagus; Adenocarcinoma of the Stomach; Adenocarcinoma - GEJ; Squamous Cell Car. - Esophagus
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Baseline tumour biopsy, biopsy at progression. Research blood, saliva stool as appropriate.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early stage curative disease
  Interventions: Diagnostic Test: biopsy
- Locally advanced or metastatic disease
  Interventions: Diagnostic Test: biopsy

INTERVENTIONS:
Diagnostic Test: biopsy — Baseline biopsy and biological specimens

SUMMARY:
A prospective translational tissue collection study to identify biomarkers predictive of treatment response/resistance and biomarkers of prognostic value from a series of patients who are investigated for and diagnosed with early or advanced gastric/junctional or oesophageal cancer (oesophagogastric cancer) at The Royal Marsden Hospital.

DETAILED DESCRIPTION:
Tissue samples and biological specimens (which may include blood, stool, saliva) from patients with a suspected/confirmed oesophagogastric cancer (OGC) at The Royal Marsden NHS Foundation Trust over the study period will be collected and stored on behalf of The Royal Marsden NHS Foundation Trust. Molecular analyses including, but not limited to, miRNA analysis, DNA and RNA sequencing, nanostring, RT-PCR and immunohistochemistry will be carried out. Stool and saliva samples may be analysed to assess the microbiota present. Molecular analyses data and microbiota data will be collated in a link-anonymised manner and correlated to clinical outcome data.

This prospective study is intended to set up a database of patients treated both for oesophageal cancer and gastric cancer with availability of annotated clinical data and tumour tissue plus biological specimens. This series will serve as a valuable platform to analyse the expression of several biomarkers of potential interest. There will also be the opportunity to assess the prognostic and predictive role of identified biomarkers in specific patient subgroups and in relation to specific treatments. Within this study, we may also hope to develop organoid and patient derived xenograft models to represent locally advanced and metastatic disease which will support future drug development. We aim to also investigate the microbiome of patients diagnosed with OGC. In addition, this database can serve as a validation cohort for the external validation of findings from other projects in OGC which are of clinical relevance. The molecular analysis plans for the study will develop as the study progresses and as new data emerges which will generate new hypotheses to investigate.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is being investigated/treated for OGC at The Royal Marsden Hospital during the study period.
2. Patient has an oesophageal/gastric mass or metastasis amenable to core needle biopsy or surgery.
3. Patient is clinically fit enough to undergo a tumour biopsy or surgery (if not already performed) according to investigator assessment and local guidelines.
4. Patient is ≥ 18 years of age.
5. Patient is able to understand the information provided within the patient information sheet and is able to provide written informed consent.
6. Patient has sufficient tissue for analysis.

Exclusion Criteria:

1. Patients who are not treated at The Royal Marsden Hospital or referring centre.
2. Patients who have a second active malignancy other than oesophageal/gastric cancer.
3. Patients who have one or more contraindications to a tumour biopsy or surgery (if not already performed) according to local guidelines.
4. Patients with an uncontrolled concomitant medical condition including, but not limited to, ongoing or active infection not amenable to standard antibiotic therapy, irreversible increased risk of bleeding which prevents biopsy as per standard procedures, or a psychiatric illness or social situation that could affect compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing endoscopy or surgery for OGC (adenocarcinoma or squamous cell carcinoma) or patients who have recently with been diagnosed with OGC and are due to start treatment. Patients will be recruited from The Royal Marsden NHS Foundation Trust. Patients will need to have sufficient tissue to be available for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
The prevalence and distribution of biomarkers potentially prognostic or predictive of treatment response/resistance in a large series of patients with OGC | 5 years

SECONDARY OUTCOMES:
Disease control rate (CR, PR and SD) in locally advanced/metastatic disease | 5 years
Duration of response (CR/PR) in locally advanced/metastatic disease | 5 years
Progression free survival (PFS) in locally advanced/metastatic disease | 5 years
Relapse free survival (RFS) in early stage curative disease | 5 years
Overall Survival (OS) according to stage of disease | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr Avani Athauda, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust - London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided